CLINICAL TRIAL: NCT06518811
Title: Özel Gereksinimli Çocuğu Olan Ebeveynlerde Telerehabilitasyon Uygulamasının Ağrı, Yetersizlik, Anksiyete ve Depresyon, Fiziksel Aktivite Seviyesi ve Yaşam Kalitesi Üzerine Etkisi
Brief Title: The Effect of Telerehabilitation on Pain, Physical and Biopsychosocial Factors in Parent Carers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ilke KARA (Other)
Responsible Party: Sponsor-Investigator, Ilke KARA, Co-Investigator, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: DEU-FTR-IK-03
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Muskuloskeletal Diseases
Keywords: Telerehabilitaton; Video-Based Exercises; Parent Carer

STUDY DESIGN:
Who Masked: Participant
Masking Description: Eligible individuals will be randomly allocated to either the exercise group or the control group. Participants will be blinded to their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): The asynchronous video-based telerehabilitation programme had a duration of eight weeks. The exercise group participants were instructed to perform the exercises on a regular basis, three days a week, with a time interval of 24 hours between each session. The exercises were to be performed using the instructional videos and recorded in the exercise diaries provided.
  Interventions: Other: Video-Based Exercise Programme
- Control group (No Intervention): Control group participants were informed about the benefits of ergonomic training for activities of daily living. Also handbooks containing the same information were distributed.

INTERVENTIONS:
Other: Video-Based Exercise Programme — The asynchronous video-based telerehabilitation programme had a duration of eight weeks. The participants were instructed to perform the exercises on a regular basis, three days a week, with a time interval of 24 hours between each session. The exercises were to be performed using the instructional videos and recorded in the exercise diaries provided. The participants were used exercise balls and resistance bands distributed by the researchers according to exercise programme.
  Arms: Exercise group

SUMMARY:
This study aimed to investigate the effects of asynchronous video-based exercises on pain, disability, anxiety, care burden and quality of life in parent carers of children with special needs.

DETAILED DESCRIPTION:
This study aimed to investigate the effects of asynchronous video-based exercises on pain, disability, anxiety, care burden and quality of life in parent carers of children with special needs.

Parents carers were invited to participate in the study through a variety of channels, including printed posters, corporate social media posts, phone calls through local administrations and non-governmental associations. At the information meeting, the participants were informed about the benefits of ergonomic training for activities of daily living. Also handbooks containing the same information were distributed. Demographic data were collected, and questionnaires were used to assess pain, disability, physical activity levels, care burden, and quality of life.

Individuals who met the inclusion criteria were randomly assigned to either the exercise group or the control group. The exercise group was informed of the details of the study methodology, technology literacy, and tablet usage. In order to ascertain an appropriate exercise programme for each individual, the researchers identified musculoskeletal problems of participants. The exercise programme comprised videos of relaxation, postural control and muscle strengthening exercises, which were recorded by research team and uploaded to the tablets. Subsequently, the participants were informed of the safety precautions during the exercise programme at home and the ergonomic placement of the tablets.

The eight-week exercise programme required participants to perform the exercises on a regular basis, three times per week, with the assistance of guided videos. Additionally, they were required to record their performance in written exercise diaries, which were distributed to them.

Exercises also supported by online calls made by the researchers once a week. In each interview, the participants were reminded of the next scheduled online interview activity. At the end of the eight-week, final evaluations were obtained through face-to-face interviews.

ELIGIBILITY:
Inclusion Criteria:

* The individual must be the primary caregiver of a child with physical, mental, or a combination of both disabilities.
* The individual must have been in this role for a minimum of six months.
* Willing to participate in the study.
* Able to read and write in Turkish.

Exclusion Criteria:

* A clear cognitive or language disability
* A recent deterioration of family relationships or the presence of factors affecting them (separation of parents, divorce, etc.)
* A history of cardiac or pulmonary disease or diseases (uncontrolled hypertension, arrhythmia, COPD, asthma, etc.), neurological disease, orthopaedic or rheumatological disease (rheumatoid arthritis, ankylosing spondylitis, arthrosis, etc.)
* A disease that may prevent exercise or that has resulted in surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 8 weeks
  Pain intensity is measured using a visual analogue scale (VAS). The level of pain felt at rest and during activity is recorded on a 10-centimetre scale. A score of zero indicates no pain and '10' indicates unbearable pain.
Scandinavian Musculoskeletal Questionnaire | 8 weeks
  The Scandinavian Musculoskeletal Questionnaire was used to assess musculoskeletal problems. The questionnaire employs a pictorial representation of the body, comprising images of the neck, shoulders, back, elbows, wrists/hands, waist, hips/thighs, knees, and ankles/feet, to elicit responses pertaining to musculoskeletal complaints. For each body part, three questions are posed, even in the absence of any perceived issues. For each specified area, participants are asked whether they have experienced a physical problem in the preceding 12 months, 1 month, and in the last 7 days. They are also asked whether they have fallen behind in their academic or professional activities as a result of this problem. Each question on the questionnaire is included in the evaluation, with a value of '1' assigned to a positive response and '0' assigned to a negative response.

SECONDARY OUTCOMES:
Zarit Scale of Caregiver Burden | 8 weeks
  The level of care burden was evaluated using the Zarit Scale of Caregiver Burden. The scale comprises a total of 22 questions, including items that examine the physical, mental, social and economic aspects of the caregiver role. The scale items are scored on a four-point Likert scale, with the options "0=Never", "1=Rarely", "2=Sometimes", "3=Frequently" and "4=Almost always". The total score is obtained by summing the scores given to each item. The total score obtained from the scale is indicative of the degree of care burden. A total score of 0-20 is indicative of a 'little or no care burden', a score of 21-40 is indicative of a 'light care burden', a score of 41-60 is indicative of a 'moderate care burden', and a score of 61-88 is indicative of a 'heavy care burden'.
Neck Disability Index | 8 weeks
  The Neck Disability Index assesses the severity of neck pain, symptoms, duration and disability in the activities listed in each item. Each item has 5 options and is scored from 0 to 4 points. The total score for neck pain is 36 points. If patients do not drive, the total score is calculated using 32 points.
Oswestry Disability Index | 8 weeks
  The Oswestry Disability Index has 10 sections including pain intensity, ability to perform daily tasks, heavy lifting, walking, sitting, standing, sleeping, sexual life, social life and travel. The participant is asked to select the statement that best describes their condition from 6 options. The patient is scored on a range of 0-20 points if their daily life is minimally affected, 20-40 points if it is moderate, 40-60 points if it is severe, 60-80 points if it is completely restricted and 80-100 points if they are bedridden.
International Physical Activity Level Questionnaire-Short Form | 8 weeks
  Physical activity was assessed using the International Physical Activity Level Questionnaire-Short Form (IPAQ). It consists of seven questions and provides information on time spent in walking, moderate-intensity and vigorous-intensity activities and time spent sitting during the past week.
Adult Carer Quality of Life Questionnaire | 8 weeks
  Quality of life was assessed using the Adult Carer Quality of Life Questionnaire, a 40-item tool developed specifically for adult carers, which provides the opportunity to assess quality of life in 8 different domains: caregiving, care preferences, caregiving stress, financial issues, personal development, appreciation, caregiving ability and carer satisfaction.
Hospital Anxiety and Depression Scale | 8 weeks
  Levels of anxiety and depression were assessed using the Hospital Anxiety and Depression Scale. Out of a total of 14 questions, seven assess anxiety and seven assess depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No